CLINICAL TRIAL: NCT05172726
Title: A Phase 3 Study of Tapinarof for the Treatment of Plaque Psoriasis in Pediatric Subjects
Brief Title: Tapinarof for the Treatment of Plaque Psoriasis in Pediatric Subjects
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMVT-505-3004
Record Dates: First submitted 2021-10-28; First posted 2021-12-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; pediatric; phase 3; topical; tapinarof

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: tapinarof cream, 1%

INTERVENTIONS:
Drug: tapinarof cream, 1% — applied topically once daily

SUMMARY:
This is an open-label, multi-center, Phase 3 study to evaluate tapinarof cream, 1% in pediatric subjects with plaque psoriasis.

DETAILED DESCRIPTION:
This study is an open-label study, consisting of a 12-week primary treatment phase and an optional 40-week long-term extension phase in which all eligible subjects will receive tapinarof cream, 1% once daily. At the end of the 12-week primary treatment phase subjects will have the option to continue for 40 additional weeks of treatment. Subjects who choose not to participate in the optional 40-week long-term extension phase will complete a follow-up visit approximately one week after the end of the primary treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 2 to 17 years with clinical diagnosis of chronic plaque psoriasis and stable disease for at least 3 months prior to the baseline visit
* Subject with plaque psoriasis covering ≥ 3% of the BSA at screening and baseline
* A PGA score of ≥ 2 at screening and baseline
* Female subjects of childbearing potential who are engaging in sexual activity that could lead to pregnancy should use acceptable birth control methods
* Must not be pregnant
* Subject, subject's parent, or legal representative must be capable of giving written informed consent/assent

Exclusion Criteria:

* Psoriasis other than plaque variant
* Any sign of infection of any of the psoriatic lesions
* Immunocompromised at screening
* Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2.0x the upper limit of normal (ULN)
* Screening total bilirubin > 1.5x ULN
* Current or chronic history of liver disease
* Current or history of cancer within 5 years except for adequately treated cutaneous basal cell carcinoma, squamous cell carcinoma or carcinoma in situ of the cervix
* Major surgery within 8 weeks prior to baseline or has a major surgery planned during the study
* Known history of clinically significant drug or alcohol abuse in the last year prior to baseline
* Use of any prohibited medication or procedure within the indicated period before the baseline visit until the completion of the study completion or study discontinuation
* History of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion may interfere with the subject's participation in the study, interpretation of results, safety of the subject or ability to understand and give informed consent
* Pregnant or lactating females.
* History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation
* Previous known participation in a clinical study with tapinarof (previously known as GSK2894512 and WBI-1001)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening up to Week 53
  Incidence, frequency, and duration of treatment emergent AEs and SAEs
Number of subjects with clinically significant laboratory test abnormalities | Screening up to Week 53
Number of subjects with clinically significant vital signs abnormalities | Screening up to Week 53
Investigator-Assessed Local Tolerability Scale (LTS) Scores | Baseline up to Week 52
  Local Tolerability Scale (LTS) is a clinical tool for assessing the presence and overall degree of irritation at the application sites, according to a 5-point scale (0-4). Higher LTS scores represent more severe irritation.
Subject (or Caregiver)-Assessed Local Tolerability Scale (LTS) | Baseline up to Week 52
  Local Tolerability Scale (LTS) is a clinical tool for assessing the presence and overall degree of irritation at the application sites, according to a 5-point scale (0-4). Higher LTS scores represent more severe irritation.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Detectable Time-Point (AUC0-t) of tapinarof cream, 1%. | Week 4 and Week 12
  Area under the plasma concentration-time curve from time zero to the last quantifiable time point.
Maximum Plasma Concentration (Cmax) of tapinarof cream, 1%. | Week 4 and Week 12
  Maximum observed plasma concentration (Cmax).
Time to Maximum Plasma Concentration (tmax) of tapinarof cream, 1%. | Week 4 and Week 12
  Time to maximum observed plasma concentration obtained directly from the observed concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead Late-Stage Clinical Development, Study Director — Organon and Co
Locations (19):
- United States (12):
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - RM Medical Research, Miami Lakes, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Options Research Group, West Lafayette, Indiana
  - Wright State Physicians Pharmacology Translational Unit, Fairborn, Ohio
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (7):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Rejuvenation Laser Dermatology Clinics, Edmonton, Alberta
  - Skincare Studio INC, St. John's, Newfoundland and Labrador
  - Lynderm Research Inc., Markham, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - Whitby Health Centre Dermatology Trials, Whitby, Ontario
  - Innovaderm Research, Inc., Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No